CLINICAL TRIAL: NCT04570163
Title: Berlin Registry of Right Heart Interventions
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Henryk Dreger, Professor, Charite University, Berlin, Germany
Other Study IDs: EA1/043/20
Record Dates: First submitted 2020-09-20; First posted 2020-09-30 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Tricuspid Regurgitation; Pulmonary Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Pulmonary Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Interventional therapy mainly of tricuspid regurgitation (TriClip, Cardioband) — Catheter-based therapy of valve diseases of the right heart with various devices (e. g. TriClip, Cardioband).

SUMMARY:
The present study evaluates patients after interventional therapy of valvular diseases of the right heart. Follow-up examinations include medical history taking, laboratory measurements and an echo. The aim is to assess the different interventional therapies and their impact on patient's outcome.

DETAILED DESCRIPTION:
The subject of the study is to register interventional therapies of right heart diseases (such as "cardioband" and "edge-to-edge" techniques of the tricuspid valve) performed in Berlin/ Brandenburg (primarily at the Charité, Universitätsmedizin Berlin). Based on the development and the increasing use of interventional therapies in tricuspid and pulmonary valve diseases, the impact on the patients' symptoms and life expectancy after interventions will be investigated. The aim is to identify patient subgroups that benefit the most.

Primary endpoints: Total mortality, cardiovascular mortality, heart failure hospitalization.

Secondary endpoints: NYHA class, NTproBNP, liver and kidney function (laboratory measurements), valve function, cardiac function, and cardiac morphology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with planned or recent valve interventions of the right heart (tricuspid regurgitation/ stenosis, pulmonary regurgitation/ stenosis)
* >18 years
* Written, documented consent

Exclusion Criteria:

* Patients in care or unable to consent
* Patients who are unable to comply with follow-up examinations
* Patients who are detained in an institution

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients after interventional therapy of valvular diseases of the right heart (such as "cardioband" and "edge-to-edge" techniques of the tricuspid valve) performed in Berlin/ Brandenburg (primarily at the Charité, Universitätsmedizin Berlin).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall mortality | 2 months after intervention
  Number of deceased participants after 2 months after intervention
Cardiovascular mortality | 2 months after intervention
  Number of deceased participants after 2 months after intervention (cardiovascular cause of mortality)
Unscheduled hospitalization for heart failure progression | 2 months after intervention
  Number of participants with unscheduled hospitalization for heart failure progression after 2 months after intervention

SECONDARY OUTCOMES:
NYHA class | 2 months after intervention
  New York Heart Association (NYHA) class (to rate dyspnea in heart failure patients)
NTproBNP | 2 months after intervention
  Laboratory measurement of NTproBNP 2 months after intervention
valve function | 2 months after intervention
  Echocardiographic quantification of valve function (proximal isovelocity surface area [PISA] method, effective regurgitant orifice [ERO], vena contracta [VC]) after 2 months after intervention
liver function | 2 months after intervention
  Laboratory measurement of bilirubin 2 months after intervention
kidney function | 2 months after intervention
  Laboratory measurement of creatinine 2 months after intervention
cardiac function | 2 months after intervention
  Echocardiographic measurement of cardiac function (left ventricular ejection fraction, tricuspid anular plane systolic excursion) after 2 months after intervention
cardiac morphology | 2 months after intervention
  Echocardiographic measurement of cardiac morphology (right ventricular and right atrial diameter) after 2 months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
As part of the expected publications, it is planned to provide data of the study participants and more detailed information on inclusion and exclusion criteria (study protocol).